CLINICAL TRIAL: NCT00591422
Title: Phase I Study of Oral Darinaparsin (ZIO-101-C) in Advanced Solid Tumors and Non-Hodgkin's Lymphomas
Brief Title: Phase I Study of Oral Darinaparsin (ZIO-101-C)in Advanced Solid Tumors and Non-Hodgkin's Lymphomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGC1001
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancer
Keywords: Arsenic; Cancer
MeSH Terms: conditions — Neoplasms | interventions — darinaparsin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: ZIO-101-C (Darinaparsin)

INTERVENTIONS:
Drug: ZIO-101-C (Darinaparsin) — Capsule, Dose escalation study from 100 mg to 1000 mg (or Maximum Tolerated Dose). 3 times weekly (>36 hours between doses) for 3 weeks with 1 week rest.
  Other Names: ZIO-101-C

SUMMARY:
The study of Dariniparsin (ZIO-101-C) in Advanced Solid Tumors and Non-Hodgkin's Lymphomas

ELIGIBILITY:
Inclusion Criteria

1. Patients with non-Hodgkin's Lymphomas that are refractory to standard therapies for their condition.(As of protocol amendment 6.0 dated 8/26/2009)
2. Men and women of ≥ 18 years of age.
3. ECOG performance score ≤ 2 (see Appendix 4).
4. Eligible subjects with lymphomas must have measurable disease as defined by the revised International Working Group response criteria (Appendix 7)
5. Life expectancy ≥ 12 weeks.
6. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements, to be conducted <2 weeks prior to Baseline:

   * Creatinine ≤ 2X upper limit of normal (ULN) OR a calculated creatinine clearance ≥ 50 cc/min
   * Total bilirubin ≤ 2X ULN
   * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 3X ULN
   * Granulocytes in peripheral blood ≥1 x 109/L, hemoglobin ≥8.5 g/dL, and platelets ≥50,000 /µL
7. Written informed consent in compliance with ZIOPHARM policies and the Human Investigation Review Committee (IEC/IRB) having jurisdiction over the site.

Exclusion Criteria

1. New York Heart Association (NYHA) functional class ≥3 myocardial infarction (see Appendix 5) within 6 months.
2. Uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation; a QTc ≥450 msec; or a ≥Grade 2 atrioventricular (AV) block or left bundle branch block (LBBB); or documented history of prolonged QTc.
3. Pregnant and/or lactating female. (Women of childbearing age must use effective contraception from Screening through the duration of Study participation.)
4. Uncontrolled systemic infection (documented with microbiological studies).
5. Metastatic brain or meningeal tumors.
6. Patients with seizure disorder requiring medication (such as anti-epileptics).
7. History of confusion or dementia or neurological condition that could mask a potential adverse response to Study Drug which may include transient ischemic attack, Parkinson's disease, thrombotic or hemorrhagic stroke, Alzheimers, and other neurological disorders.
8. Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of Study entry (mitomycin C or nitrosureas should not be given within 6 weeks of Study entry).
9. Radiotherapy during study or within 3 weeks of Study entry.
10. Surgery within 4 weeks of start of Study Drug.
11. Investigational drug therapy outside of this trial during or within 4 weeks of Study entry.
12. History of invasive second primary malignancy diagnosed within the previous 3 years except for Stage I endometrial/cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer.
13. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of Study results.
14. Any condition that is unstable or could jeopardize the safety of the patient and his/her compliance in the Study.
15. Arsenic allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-08; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Toxicities | 6 months

SECONDARY OUTCOMES:
pharmacokinetics | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lewis, MD, PhD, Study Director — Alaunos Therapeutics
Locations (3):
- United States (3):
  - Ocoee, Florida
  - Dallas, Texas
  - Norfolk, Virginia